CLINICAL TRIAL: NCT00680160
Title: An Open-label, Multiple-dose Study Of The Absorption And Systemic Pharmacokinetics Of An2690 Applied As A 7.5% Solution To All Toenails Of Adult Patients With Moderate To Severe Onychomycosis
Brief Title: Absorption and Systemic Study of AN2690 in Patients With Moderate to Severe Onychomycosis (ADME I)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: AN2690-ONYC-202; C3371013 (Other: Alias Study Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis | interventions — tavaborole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AN2690 — AN2690 7.5% Solution, once daily for 28 days

SUMMARY:
The purpose of the study is to determine the absorption, systemic pharmacokinetics and accumulation in the nail of AN2690 during a 28 day period of daily application of a 7.5% solution of AN2690 to all 10 toenails of up to 25 otherwise healthy adult patients with onychomycosis.

DETAILED DESCRIPTION:
For this study, the case definition of onychomycosis included moderate to severe distal subungual onychomycosis including subjects with evidence of subungual dermatophytoma or yellow spikes, lateral and proximal onychomycosis and severely dystrophic nail plates. Subjects with only superficial white onychomycosis were excluded. Confirmation of the clinical diagnosis of onychomycosis of at least one great toenail included a positive KOH wet mount.

ELIGIBILITY:
Inclusion Criteria:

* A witnessed, signed informed consent approved by Institutional Review Board
* Male or female of any race at least 18 years of age but not older than 65 years of age at the time of screening
* Body Mass Index between 18.5 and 35, inclusive
* Onychomycosis involving > 80% of both great toenails, as determined by visual inspection after the nail has been trimmed
* Each great toenail possess a combined thickness of the nail plate and nail bed > 3 mm
* At least six additional toenails with clinical diagnosis of onychomycosis
* A positive KOH wet mount for at least one great toenail
* If subject is a female of childbearing potential, must be using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices) during the study
* Considered reliable and capable of understanding his/her responsibility and role in the study

Exclusion Criteria:

* History of allergy to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure
* Clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his/her safety
* Diabetes mellitus requiring treatment other than diet and exercise
* Unwilling to refrain from the use of nail cosmetics such as clear and or colored nail lacquers from the screening visit until the end of the study
* Nursing, pregnant or planning to become pregnant during the study
* Has not undergone the specified washout period(s) for the following topical preparations or does the subject require the concurrent use of any of the following topical medications:

  1. Topical antifungal applied to the feet (does not include antifungals for treatment of T. pedis during the study: 4 weeks
  2. Anti-inflammatories, corticosteroids, topical immunomodulators: 2 weeks
* Has not undergone the specified washout period(s) for the following systemic medications or does the subject require the concurrent use of any of the following systemic medications:

  1. Corticosteroids (including intramuscular injections): 2 weeks
  2. Antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophyte: 24 weeks
  3. Systemic immunomodulators: 4 weeks
* Received treatment of any type for cancer within the last 6 months
* History of any significant internal disease
* Nail or anatomic abnormalities of the toe, e.g., genetic nail disorders, primentary disorders, onychogryphosis, trauma to the nail(s) to be treated
* AIDS or AIDS related complex
* History of street drug or alcohol abuse
* Donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation
* Donated plasma during the two week period preceding study initiation
* Participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-04-30 (Actual); Primary Completion 2007-05-09 (Actual); Study Completion 2007-05-09 (Actual)

PRIMARY OUTCOMES:
Efficacy measures of linear toenail growth, fungal culture results, KOH results, and clear toenail | Days 0, 14, 28, 42, 84, 120, 150, 180, 240, 300, and 360

SECONDARY OUTCOMES:
Safety and tolerance assessed by application site reactions, adverse events, laboratory tests, vital signs, physical examinations, and 12-lead EKG | Days 0-28, 42, 84, 120, 150, 180, 240, 300, and 360

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- J&S Studies, Bryan, Texas, United States